CLINICAL TRIAL: NCT03537521
Title: Prospective, Observational, Non-interventional Open-Label, International, Multicenter Registry Regarding the Management of Severe Bleeding and/or Urgent Interventions During Treatment With Direct Oral Anticoagulants or Vitamin K Antagonists
Brief Title: Reversal Agent Use in Patients Treated With Direct Oral Anticoagulants or Vitamin K Antagonists (RADOA). Focus on New Antidots
Status: Withdrawn | Type: Observational
Why Stopped: due to corona pandemic crisis
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Sponsor
Other Study IDs: RADOA.DOT
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Severe Bleeding; Urgent Surgery
Keywords: severe bleeding; dabigatran; rivaroxaban; apixaban; edoxaban; PCC; aPCC; rVIIa; hemodialysis; antidots; idarucizumab; urgent surgery; andexanet alpha
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — If possible, left-over from plasma samples ("retention sample") should be used to perform further analyses as drug concentrations. Retention samples of very low volume would suffice for HPLC (information on collection method needed) to assess plasma concentrations of anticoagulants in these patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DOA: N= 130 patients treated with direct oral anticoagulants (DOAC) with acute bleeding N= 65 patients treated with direct oral anticoagulants (DOAC) with urgent surgical intervention
  Interventions: Procedure: Urgent surgery which can not be postponed to the next 24 hrs
- VKA: N= 130 patients treated with vitamin K antagonists (VKA) with acute bleeding N= 65 patients treated with vitamin K antagonists (VKA) with urgent surgical intervention
  Interventions: Procedure: Urgent surgery which can not be postponed to the next 24 hrs

INTERVENTIONS:
Procedure: Urgent surgery which can not be postponed to the next 24 hrs — The urgent surgical intervention is not part of the registry protocol. The intervention is the acute event that leads to enrollment in the registry. It might be e.g. the surgical treatment of a trauma, fall, acute abdomen, appendicitis or anything else.

SUMMARY:
Patients treated with Vitamin K antagonists (VKA) or direct oral anticoagulants as Rivaroxaban, Apixaban, Edoxaban or Dabigatran, who experience severe bleeding and/or need urgent interventions/operations that cannot wait are included in this registry, or during emergency operations

DETAILED DESCRIPTION:
The Registry will offer the opportunity to evaluate the effects of reversal agents as PCC, aPCC, rVIIa, specific antidots in patients needing urgent interventions/operations or in severe bleeding patients treated with oral anticoagulants.

By collecting case reports from several university hospitals and clinics, different treatment strategies in clinical practice will be observed and evaluated, and may serve as a comprehensive information resource for the safe management with DOA, but also with the long-term anticoagulation based on coumarin derivatives in the near future.

The current objective of this registry is to:

1. Document the clinical course and outcome of various clinical bleeding events associated with DOA or VKA in patients with severe life-threatening bleeding making intervention necessary
2. Document the clinical course and outcome of urgent surgical interventions within 24 hours after admission in patients under DOA or VKA treatment.
3. Characterisation of therapeutic strategies in stopping acute life-threatening bleeding including following agents and methods:

   1. blood transfusion,
   2. platelet concentrates
   3. reversal agents [e.g. vitamin K, prothrombin complex concentrate (PCC), activated PCC (aPCC), activated factor VII (aVII), fibrinogen concentrate, fresh frozen plasma (FFP)]
   4. specific antidots, e.g. idarucizumab, Andexanet alpha
   5. haemodialysis
   6. desmopressin
   7. tranexamic acid
   8. no specific treatment in respect to the above mentioned treatments (e.g. stop of medication and waiting until anticoagulant effect of DOA is decreased).

ELIGIBILITY:
Inclusion Criteria:

Group a) Bleeding patients:

* Anticoagulated patients with DOA or VKA with clinically overt major bleeding according to a specified ISTH definition for non-surgical patients:
* Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome
* Bleeding causing a fall in hemoglobin level of 2 g L-1 (1.24 mmol L-1 ) or more leading to transfusion of two or more units of whole blood or red cells.

OR

Group b) Acute surgical need patients

* treated with DOA or VKA and who need urgent operation which cannot wait (< 24 h after last intake of drug)
* with or without reversal agent use (e.g. PCC, aPCC, rVIIa) (and/or haemodialysis for dabigatran)
* provides informed consent after the acute event

Exclusion Criteria for Group a and b:

* Conscious patient by him-/ herself or his/ her available legal representative does not agree with inclusion in the registry
* Age < 18 years
* Concomitant participation in an interventional trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Expected number of patients estimated by study duration
  N= 130 patients treated with direct oral anticoagulants (DOA) with acute bleeding N= 130 treated with vitamin K antagonists (VKA) with acute bleeding
  N= 65 patients treated with direct oral anticoagulants (DOA) with urgent surgical intervention N= 65 patients treated with vitamin K antagonists (VKA) with urgent surgical intervention
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality up to 30 days after admission | up to 30 days after hospital admission
  Death rate (number of deaths)

SECONDARY OUTCOMES:
Stop of bleeding defined according to the treating physicians | up to 30 days after hospital admission
  Decission according to the treating physicians
Fatality rate caused by unstoppable bleeding | up to 30 days after hospital admission
  Death rate (number of deaths)
Use versus no use of reversal agents - difference in outcome? | up to 30 days after hospital admission
  documentation of use of reversal agents in eCRF
Definition of supportive measures being effective in stopping bleeding | up to 30 days after hospital admission
  documentation of supportive measures in eCRF
Effectiveness of dialysis vs. no dialysis in case of dabigatran accumulation associated with bleeding | up to 30 days after hospital admission
  time frame until stop of bleeding
Causality assessment: Relation of SAE to anticoagulant medication | up to 30 days after hospital admission
  Decission according to the treating physicians
Blood loss, number of transfusions necessary | up to 30 days after hospital admission
  documentation of supportive measures in eCRF
Satisfaction of surgeon during and after surgery concerning bleeding | up to 30 days after hospital admission
  Decission according to the treating physicians
Use versus no use of reversal agents - difference in blood loss and number of transfusions | up to 30 days after hospital admission
  documentation of supportive measures in eCRF
Delay in performance of surgery due to anticoagulation | up to 30 days after hospital admission
  time Frame documented in eCRF

CONTACTS AND LOCATIONS:
Overall Officials: Edelgard Lindhoff-Last, Prof., Principal Investigator — CCB Studienzentrum GmbH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindhoff-Last E, Herrmann E, Lindau S, Konstantinides S, Grottke O, Nowak-Goettl U, Lucks J, Zydek B, Heymann CV, Birschmann I, Sumnig A, Beyer-Westendorf J, Schellong S, Meybohm P, Greinacher A. Severe Hemorrhage Associated With Oral Anticoagulants. Dtsch Arztebl Int. 2020 May 1;117(18):312-319. doi: 10.3238/arztebl.2020.0312. PMID 32605708